CLINICAL TRIAL: NCT06977113
Title: The Effect of Maternal High Fibre and Fermented Food Rich Diet on Breastfed Infant Gut Microbiome: A Randomised Controlled Trial
Brief Title: Maternal High Fibre Fermented Diet Effect on Breastfed Infant Gut Microbiome
Acronym: MumBabyGut
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Ada Garcia, Senior Lecturer in Public Health Nutrition, School of Medicine, Dentistry & Nursing, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 200240089
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Mothers; Healthy Infants
Keywords: maternal diet; breast milk; infant gut microbiome; dietary fibre; fermented food; human milk oligosccharide; short chain fatty acids; gut microbiota; Exclusive breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study intervention, which involves the use of whole foods that cannot be effectively concealed, both study researchers and participants will be unblinded to group allocation during the intervention. However, to minimize bias and ensure objective evaluation, study researchers involved in data analysis will be blinded to the group assignments throughout the analysis process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fibre Fermented Food Diet (Experimental): Participants in this arm will be assigned to consume specific foods that are high in fibre and fermented products (25 g fibre/day) in addition to their usual diet for two weeks. These foods include oatcakes or oat porridge, shredded wheat cereal biscuits, a high-fibre bar, yogurt and kefir, as well as two of the following: hummus, lentil soup, or baked beans. These foods will only be consumed by the mothers and they will be instructed to eat specific portion sizes of each food item per day. Researchers will provide participants with a dietary checklist to help them record their daily intake of the study foods for the 2-week study period. Participants will be asked to avoid consuming probiotic and prebiotic supplements during the 2-week study intervention.
  Interventions: Other: High Fibre Fermented Food Diet
- Control Habitual Diet (Other): Participants assigned to the control group will maintain their habitual diet, and they will not be given any of the study foods. Participants will be asked to avoid consuming probiotic and prebiotic supplements throughout the 2-week study period. The population average fibre intake for women in Scotland is 16 g/day (The Scottish Health Survey 2021).
  Interventions: Other: Control Habitual Diet

INTERVENTIONS:
Other: High Fibre Fermented Food Diet — Participants will be provided with and asked to consume specific foods high in various types of fibre to promote a variety of substrates for gut bacteria including inulin, galactooligosaccharides (GOS), and β-glucan. Participants will also be asked to consume 2 fermented items, yogurt and kefir. Study foods will be commercially available including a high-fibre bar made from chicory-derived inulin (1 bar of 35 g/d), oat-containing cakes (4 oatcakes of 35 g/d) or oat porridge (1 sachet of 38.5 g/d), shredded wheat cereal biscuits (2 biscuits of 45 g/d), hummus (½ pot of 100 g/d), and/or baked beans (½ can of 100 g/d) or lentil soup (1 can of 400 g/d), and low fat yogurt (1/3 pot of 150 g/d) and kefir (½ bottle of 250 ml/d). The total amount of fibre study foods will provide is approximately 25 g/day which will be consumed in addition to the habitual diet. The total amount of fibre will be expected to reach the 30 g/day recommendation and will range between 25 - 40 g/day.
  Arms: High Fibre Fermented Food Diet
Other: Control Habitual Diet — Participants will follow their habitual diet and will not consume any of the study foods (i.e., high-fibre fermented foods). The population average fibre intake for women in Scotland is 16 g/day (The Scottish Health Survey 2021).
  Arms: Control Habitual Diet

SUMMARY:
Breastfeeding is recommended for babies from birth to six months old because breast milk provides all the nutrients babies need for growth and development. Breast milk contains sugars called oligosaccharides, which support the development of a healthy gut in babies. The foods that breastfeeding mothers eat might influence the sugars in their breast milk and the natural, friendly bacteria inside their babies' gut-called the gut microbiota-which are important for overall health. Fibre-rich foods like fruits, vegetables, whole grains, beans, and nuts, as well as fermented foods like yogurt and milk kefir, support a healthy gut.

The main aim of this study is to find out whether eating foods rich in fibre and fermented foods by breastfeeding mothers can affect the bacteria residing in the gut of their breastfed babies. The study will also explore how this diet affects the mother's gut microbiota, breast milk composition, and gastrointestinal (GI) symptoms for both mothers and babies.

The main question of the study is: Does a 2-week diet high in fibre and fermented foods consumed by breastfeeding mothers affect the gut microbiota of their breastfed babies aged 2 to 5 months, compared to mothers following their habitual diet?

Participants will:

* Be randomly assigned to one of two groups: (1) one group will follow a specific diet high in fibre and fermented foods (25 g of fibre/day + 3 servings of fermented foods/day) in addition to their habitual diet, or (2) the second group will continue with their habitual diet (no specific foods will be provided) (16 g of fibre/day).
* Attend a single study visit at the study location.
* Provide body measurements (weight and height) of mothers and babies at the. study visit, and provide weight only during each home visit.
* Complete gut health questionnaires for both mothers and babies twice during the study.
* Complete two sets of 3-day, 24-hour dietary recalls during the study.
* Provide stool samples (3 from babies and 2 from mothers) and 2 breast milk samples.

Researchers will then compare the stool samples from both mothers and babies to see whether the specific diet makes any difference to the gut microbiota.

DETAILED DESCRIPTION:
Study duration:

The study will span a total of three weeks, comprising a one-week run-in period followed by a two-week intervention period.

Recruitment:

Healthy, exclusively breastfeeding women aged over 18 years and their healthy infants aged between 2 to 5 months will be recruited from the general population residing in the Glasgow & Clyde area of Scotland. The study will be advertised using posters distributed through various channels, including word of mouth, breastfeeding support groups, schemes, venues, and organisations, as well as social media platforms. Researchers will screen potential participants for eligibility and only recruit healthy participants (i.e., healthy mothers and infants). Eligible participants will be invited to attend a one-hour study visit at the researchers' metabolic facilities for further screening.

Study visit:

Researchers will recheck participants' eligibility, reiterate the study purpose and requirements, and address any questions or concerns participants may have. If participants choose to proceed, they will be asked to sign a consent form but will be made aware that they can withdraw at any time. Each participant will be assigned a unique study identification number for anonymisation purposes, and the data retention policy will be explained up to the point of withdrawal.

Sociodemographic information will be collected using a questionnaire, and anthropometric measurements will be assessed for both mothers and infants. Maternal body weight (in kg) in light clothing and barefoot will be measured using an electronic scale (TANITA), and maternal height (in cm) using a stadiometer. Maternal BMI (in kg/m²) will be calculated. The infant's weight will be measured without a nappy (diaper). Infant body weight (in kg) and length (in cm) will be obtained using a baby scale and infantometer (SECA), with the assistance of the mother or caregiver.

The specific procedures for the study protocol will be explained to participants. Researchers will provide the necessary kits and instructions for sample collection (stool and breast milk). Three home visits will be scheduled, during which researchers will:

* Collect stool and breast milk samples
* Provide new collection kits
* Collect gastrointestinal (GI) paper questionnaires
* Measure the mother's and baby's weights

Post study visit:

After the study visit, participants will begin a 7-day run-in (baseline) period, during which they will:

* Follow their normal habitual diet
* Provide initial stool and breast milk samples
* Complete dietary assessments and GI questionnaires

The tools used include:

* A 3-day multiple-pass 24-hour dietary recall
* The Gastrointestinal Symptom Rating Scale (GSRS) for mothers
* The Infant Gastrointestinal Symptom Questionnaire (IGSQ) for infants

After the run-in period and collection of baseline data, participants will be randomly assigned to one of two groups:

1. Intervention group: High-fibre, fermented food-rich diet (25 g of fibre/day + 3 servings of fermented foods/day) in addition to their habitual diet
2. Control group: Habitual diet (approximately 16 g of fibre/day)

The high-fibre fermented foods will be commercially available from local grocery shops and delivered to participants' homes. Only mothers will consume the study foods; no interventions will be administered to the infants.

Researchers will follow up with participants via mobile phone to monitor deliveries, send reminders for home visits, assist with dietary recalls, and manage sample and questionnaire collection.

Data collection:

1. Questionnaires

   During the study visit, participants will complete a study visit questionnaire (covering background, dietary and pregnancy and birth information)

   After the study visit, participants will complete 3-day multiple-pass 24-hour dietary recalls at two time points - at baseline (study week 1) and at the last week of study intervention (study week 3)

   Participants will complete GSRS and IGSQ at two time points - at baseline (study week 1) and after the last week of study intervention (study week 3)
2. Biological samples

   Participants will collect biological samples, including mother's stool and breast milk, at two time points - before and after study intervention (at study week 1 and after study week 3)

   Infant's stool will be collected from nappies at three time points - before and after study intervention (at study week 1 and after study week 3) and halfway through the study (between study week 2 and week 3)

   Participants will be provided with special kits and written instructions for sample collection at home. Once samples are ready, participants will be instructed to contact the research team promptly for collection and handling.
3. Body measurements

During the study visit, mother's weight, height and body composition, and baby's weight and length will be measured. The study researcher will take the baby's measurements with the assistance of the mother or caregiver and without the nappies.

After the study visit, the study researcher will obtain the mother's and the baby's body weight at each sampling visit (or home visit), at baseline (study week 1), halfway through the study (between study week 2 and week 3), and after the last week of study intervention (study week 3).

Dietary compliance:

Fibre contents in maternal stool samples will be measured to monitor for their dietary compliance to the study intervention.

Sample size:

The sample size was calculated based on the primary outcome, which is infant faecal acetate, the predominant short chain fatty acid (SCFA) and the one expected to be affected by an increase in bifidobacteria. Based on previous randomised controlled trials, recruiting 52 mother-infant pairs would provide a power of 80% (p=0.05) to detect a significant mean change in faecal acetate of 60 μmol/g in the infant's stool (SD: 75 μmol/g). Accounting for an approximate 10% dropout rate, recruiting 56 mother-infant pairs (28 per study group) would ensure adequate power for this study.

Reimbursement:

After the completion of the study, participants will receive a gift voucher as a gesture of appreciation for their time and effort in the study. Also, participants will be reimbursed for public transport expenses to the lab.

ELIGIBILITY:
Inclusion Criteria:

* Healthy breastfeeding women aged 18 years old and older.
* Healthy singleton full-term infants (girls and boys) aged between 2 and 5 months old and who are exclusively breastfed.
* Not using lifelong medications and antibiotics in the past 12 weeks prior to the study.
* Not using prebiotic or probiotic supplements in the past 4 weeks prior to the study.
* No serious problems preventing participants from breastfeeding their babies.
* No food allergies or intolerances.
* No chronic conditions like diabetes, cancer, heart disease, bowel disorders, eating disorders, or any illness requiring regular medical care or lifelong medication.
* No history of complications during pregnancy (e.g., preeclampsia and gestational diabetes).

Exclusion Criteria:

* Expecting two or more children (i.e., multiple births; twins, triplets).
* Not exclusively breastfeeding their infants (i.e., introduced formula or solids) or having medical conditions known to contraindicate breastfeeding (e.g., classic galactosemia, human immunodeficiency virus (HIV-virus) infection, untreated tuberculosis (TB)).
* Preterm birth.
* Clinically diagnosed with chronic medical conditions (e.g., type 1 and type 2 diabetes mellitus, cancer, cardiovascular diseases, and mental illnesses).
* Medical conditions affecting gastric digestion or absorption (e.g., inflammatory bowel diseases (IBD), and irritable bowel syndrome (IBS)).
* Conditions interfering with intervention intake (e.g., celiac disease, gluten hypersensitivity or lactose intolerance).
* History of gestational complications.
* Use of antibiotics in the past 12 weeks prior to the study.
* Use of prebiotic or probiotic supplements in the past 4 weeks prior to the study.
* Following exclusionary or restrictive diets (e.g., gluten-free, or weight loss).

Ages: 2 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota and Short Chain Fatty Acids of Breastfed Infants after 2-week Dietary Intervention | From enrolment to the end of intervention at 3 weeks
  The primary objective is to evaluate whether the maternal 2-week diet rich in fibre and fermented foods alters the composition of microbiota and short chain fatty acid (SCFA) level in the gut of breastfed infants. Microbiota composition will be assessed, following stool DNA extraction, through 16S rRNA amplicon sequencing and quantitative polymerase chain reaction (qPCR). SCFA will be quantified using gas chromatography (GC) and potentially other microbial derived metabolites will be measured using other analytical techniques.

SECONDARY OUTCOMES:
Maternal Gut Microbiota and Microbial Metabolites and Breast Milk Composition | From enrolment to the end of intervention at 3 weeks
  Microbiota composition will be assessed, following stool DNA extraction, through 16S rRNA amplicon sequencing and quantitative polymerase chain reaction (qPCR). Microbial activity will be assessed by quantifying short chain fatty acids (SCFA) using gas chromatography (GC) and other microbial-derived metabolites will be measured using other analytical techniques. Breast milk samples will be analysed for human milk oligosaccharides (HMOs) profiles using high performance liquid chromatography with fluorescence detection (HPLC-FLD) or high performance liquid chromatography with ultraviolet detection (HPLC-UV). Measurement of excreted fibre in stools will also be measured using the Association of Official Analytical Chemists method.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition, School of Medicine, University of Glasgow, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study will be published in scientific peer-reviewed journal when is completed.